CLINICAL TRIAL: NCT04429984
Title: A Post Marketing Surveillance (PMS) Study for VPRIV (Velaglucerase Alfa) in India
Brief Title: Post Marketing Surveillance (PMS) Study for Velaglucerase Alfa (VPRIV) in India
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP669-406
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VPRIV: All Participants: Participants with type 1 Gaucher disease who as part of standard or routine clinical practice, have already received VPRIV retrospectively and will further receive VPRIV therapy according to the investigator's judgment for approximately 12 months will be observed prospectively in this PMS study.

SUMMARY:
The main aim of this study is to measure the safety and to find out the effects of VPRIV in participants with Gaucher disease using both retrospective and prospective data when used in the post-marketing setting and to collect genetic mutation data from participants with Gaucher disease.

This study is about collecting data available in the participant's medical record as well as data from each participant's ongoing treatment. No study medicines will be provided to participants in this study.

When the participants start the study, they will visit the study clinic close to approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 1 Gaucher disease prescribed VPRIV according to the investigator's judgment and current Indian Prescribing information (PI) are eligible for this study.
* Participants or legally authorized representative must provide written informed consent to participate.

Exclusion Criteria:

- Participants will be excluded from this study if the participant met any of the contraindications included in the current Indian PI for VPRIV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with confirmed type 1 Gaucher disease irrespective of any age or gender who have been prescribed VPRIV therapy according to the investigator's judgment will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Baseline up to approximately 12 months
  An AE is defined as any untoward medical occurrence (including a symptom or disease or an abnormal laboratory finding) in a participant or clinical investigation participants administered a medicinal product and which does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) is any event that results in: death; life-threatening event; requires inpatient hospitalization or results in prolongation of existing hospitalization; persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or a medically important event. AEs include serious adverse events, unexpected AEs, non-serious adverse events (AEs) will be reported using both retrospective and prospective data when used as standard clinical practice. Baseline is defined as measurement from first time participants was dosed on charitable access program (CAP).
Number of Participants With Adverse Drug Reactions (ADRs) | Baseline up to approximately 12 months
  An ADR is an AE for which there is at least a reasonable suspicion of a causal relationship between an AE and a suspected medicinal product. Number of participants with ADRs will be reported using both retrospective and prospective data when used as standard clinical practice. Baseline is defined as measurement from first time participants was dosed on CAP.

SECONDARY OUTCOMES:
Change From Baseline in Hemoglobin (Hb) Concentration Using Both Retrospective and Prospective Data | Baseline up to approximately 12 months
  Hemoglobin concentration will be assessed in participants with Gaucher disease receiving VPRIV using both retrospective and prospective data when used as standard clinical practice. Baseline is defined as measurement from first time participants was dosed on CAP.
Change From Baseline in Platelet Count Using Both Retrospective and Prospective Data | Baseline up to approximately 12 months
  Platelet count will be assessed in participants with Gaucher disease receiving VPRIV using both retrospective and prospective data when used as standard clinical practice. Baseline is defined as measurement from first time participants was dosed on CAP.
Change From Baseline in Spleen Size Using Both Retrospective and Prospective Data | Baseline up to approximately 12 months
  Spleen size will be assessed using ultrasound or Magnetic Resonance Image (MRI) in participants with Gaucher disease receiving VPRIV using both retrospective and prospective data when used as standard clinical practice. Baseline is defined as measurement from first time participants was dosed on CAP.
Change From Baseline in Liver Size Using Both Retrospective and Prospective Data | Baseline up to approximately 12 months
  Liver size will be assessed using ultrasound or MRI in participants with Gaucher disease receiving VPRIV using both retrospective and prospective data when used as standard clinical practice. Baseline is first time participants were dosed on CAP.
Treatment History Based on Previous VPRIV Treatment | At Baseline
  Presence of treatment history will be assessed using retrospective data of the previous VPRIV treatment. Baseline is first time participants were dosed on CAP.
Change From Baseline in Hemoglobin (Hb) Concentration Based on Previous VPRIV Treatment | Baseline up to approximately 12 months
  Hemoglobin concentration will be assessed using retrospective data of the previous VPRIV treatment. Baseline is first time participants were dosed on CAP.
Change From Baseline in Platelet Count Based on Previous VPRIV Treatment | Baseline up to approximately 12 months
  Platelet count data will be assessed using retrospective data of the previous VPRIV treatment. Baseline is first time participants were dosed on CAP.
Change From Baseline in Spleen Size Based on Previous VPRIV Treatment | Baseline up to approximately 12 months
  Spleen size date will be assessed using retrospective data of the previous VPRIV treatment. Baseline is first time participants were dosed on CAP.
Change From Baseline in Liver Size Based on Previous VPRIV Treatment | Baseline up to approximately 12 months
  Liver size data will be assessed using retrospective data of the previous VPRIV treatment. Baseline is first time participants were dosed on CAP.
Number of Participants With AEs and SAEs Based on Previous VPRIV Treatment | Baseline up to approximately 12 months
  An AE is defined as any untoward medical occurrence (including a symptom or disease or an abnormal laboratory finding) in a participant or clinical investigation participants administered a medicinal product and which does not necessarily have a causal relationship with the treatment. A SAE is any event that results in: death; life-threatening event; requires inpatient hospitalization or results in prolongation of existing hospitalization; persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or a medically important event. AEs include serious adverse events, unexpected AEs, non-serious AEs will be collected using retrospective data of the previous VPRIV treatment. Baseline is defined as measurement from first time participants was dosed on CAP. Data will be assessed retrospectively based on participant records.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (2):
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre (AIMS), Kochi, Kerala
  - All India Institute of Medical Sciences, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5facd21917465c002989a198